CLINICAL TRIAL: NCT03738553
Title: Multiparametric MRI for Assessing Breast Cancer Response to Anti-HER2 Therapy
Status: Active, not recruiting | Type: Observational
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Savannah Partridge, Professor, University of Washington
Other Study IDs: 7889; RG3013002 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2018-11-08; First posted 2018-11-13 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: HER2-positive Breast Cancer
MeSH Terms: interventions — Trastuzumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: MRI — Diffusion Weighted Imaging and Dynamic Contrast enhanced MRI
Drug: Trastuzumab — Single dose of Trastuzumab prior to surgery

SUMMARY:
This is a single institution, observational research study in which patients are observed using DWI/DCE MRI imaging before and after receiving neoadjuvant anti-HER2 therapy.

DETAILED DESCRIPTION:
This is not a treatment trial. Patients will be treated according to the plan developed by their medical oncologists. Only patients planning to receive anti-HER2 therapy as part of planned systemic therapy will be eligible for this imaging study. Patients and their referring oncologist will be asked to start the anti-HER2 therapy 2-3 weeks prior to surgery and after the pre-therapy MRI.

ELIGIBILITY:
Inclusion Criteria:

* Subjects at least 18 years of age.
* Have a new diagnosis of invasive breast cancer, clinical stage I - III, HER2 positive.
* Planning to undergo surgical resection plus adjuvant therapy to include an anti-HER2 agent.
* Have tissue block available for review of experimental markers.
* Be a candidate for MRI imaging.
* Be willing to comply with scheduled visits required for the trial.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Recent therapy for breast cancer prior to baseline MRI.
* Subjects may not receive other investigational agents during the study window for imaging.
* Contraindications for MRI or MRI contrast including severe claustrophobia, history of previous reaction to MRI contrast, renal disease, congestive heart failure, other significant systemic diseases or any metal in their body, including but not limited to: a brain aneurysm clip, implanted neural stimulator, implanted cardiac pacemaker or defibrillator, cochlear implant, ocular foreign body (e.g. metal shavings), other implanted medical devices: (e.g. Swan Ganz catheter), insulin pump, metal shrapnel or bullet.
* Pregnant or nursing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is not a treatment trial. Patients will be treated according to the plan developed by their medical oncologists. Only patients planning to receive anti-HER2 therapy as part of planned systemic therapy will be eligible for this imaging study. Patients and their referring oncologist will be asked to start the anti-HER2 therapy 2-3 weeks prior to surgery and after the pre-therapy MRI.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2020-09 (Actual); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Tumor infiltrating lymphocytes (TILs) | 10 years
  Determine whether early changes on MRI reflect the level of immune response (based on TILs) in the tumor as measured by histologic assessment after 1 cycle of anti-HER2 treatment

CONTACTS AND LOCATIONS:
Overall Officials: Savannah Partridge, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Seattle Cancer Care Alliance, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No